CLINICAL TRIAL: NCT06210438
Title: SHR-A1921 Combined With Bevacizumab in Triple-negative Breast Cancer With Brain Metastases：a Prospective, Single-arm, Single-center Phase II Clinical Study
Brief Title: SHR-A1921 Combined With Bevacizumab in Triple-negative Breast Cancer With Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCBM-003
Record Dates: First submitted 2024-01-04; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: TNBC; Brain Metastasis
MeSH Terms: conditions — Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1921 + Bevacizumab (Experimental)
  Interventions: Drug: SHR-A1921 + Bevacizumab

INTERVENTIONS:
Drug: SHR-A1921 + Bevacizumab — SHR-A1921 + Bevacizumab

SUMMARY:
This is a phaseⅡ, single-arm study evaluating the efficacy and safety of SHR-A1921 Combined with Bevacizumab in Triple-negative Breast Cancer with Brain Metastases

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, both genders
2. ECOG Performance Status of 0-2
3. Pathological tests confirm HR-negative/HER2-negative breast cancer；there is evidence of local recurrence or metastasis；not suitable with curative surgery or radiation therapy；HR negative is defined as: ER-negative and PR-negative, the proportion of positively stained tumor cells in all tumor cells is <10%；HER2- negative is defined as: histologically confirmed to be HER2 IHC (0) or HER2 IHC(1+) or HER2 IHC (2+) and FISH(-)
4. Must have life-expectancy of ≥ 3 months
5. MRI confirmed brain metastases, at least one intracranial parenchymal metastatic lesion with a longest diameter ≥ 1.0 cm without prior radiotherapy；
6. Intraventricular catheter shunting or mannitol、steroid hormone、anticonvulsant drug is allowed before enrollment, but the dose of drug should be stable for at least one week and the neurological symptoms are stable for ≥1 week
7. Adequate function of major organs meets the following requirements (1)Blood routine

   * ANC≥1.5×109/L；
   * PLT≥75×109/L；
   * Hb≥90 g/L(Allows blood transfusion or the use of medication to ensure that the content of hemoglobin) (2)Coagulation
   * INR≤1.5，APTT≤1.5×ULN (3)Blood biochemistry
   * TBIL≤1.5 × ULN;
   * ALT and AST≤3 × ULN (liver metastasis≤5.0 × ULN);
   * Urea nitrogen ≤ 1.5 × ULN; Cr≤1.5 × ULN or creatinine clearance ≥50 mL / min (Cockcroft-Gault formula) (4)Cardiac ultrasound
   * LVEF≥50%; (5)12-lead ECG:
   * females QTcF interval <470msec and males <450ms;
8. Willing to join the study, sign informed consent, have good compliance and cooperate with follow-up.

Exclusion Criteria:

1. Leptomeningeal or cystic metastases confirmed by MRI or lumbar puncture
2. Presence of third interstitial fluid that cannot be controlled by drainage or other methods (e.g., a large amount of pleural effusion and ascites);
3. Whole brain radiotherapy, chemotherapy, biological targeted therapy, immunotherapy, surgery or endocrine therapy within 2 weeks prior to enrolment
4. Has received prior therapy with bevacizumab and TROP-2 ADC drugs
5. Participation in any other clinical trials within 2 weeks of enrollment
6. Concurrent use of any other Anti-cancer drugs
7. Other malignancies within 5 years, except cured in-situ of uterine cervix carcinoma , skin basal cell carcinoma and squamous-cell carcinoma
8. History of heart disease: (1) Arrhythmias requiring medical treatment or clinical significance, (2) Myocardial infarction, (3) Heart failure, (4)Any heart diseases that investigator believes not suitable for this study
9. History of allergy or hypersensitivity to any of the study drugs or study drug components
10. History of immunodeficiency including HIV-positive, active hepatitis B/C, other acquired, congenital immunodeficiency disease or history of organ transplantation
11. A clear history of neurological or mental disorders, including epilepsy or dementia
12. Pregnant or breastfeeding women. Women of childbearing potential who have a positive pregnancy test or unwilling to use adequate contraception prior to enrollment and for the duration of study participation
13. According to the investigator's judgment, there is a concomitant disease that seriously endangers the safety of subjects or affects the completion of the study (including but not limited to severe hypertension, severe diabetes, active infection, thyroid disease that cannot be controlled by drugs)
14. Any condition which in the investigator's opinion makes the subjects unsuitable for the study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
CNS ORR | from enrollment to progression or death (for any reason), assessed up to 24 months
  The proportion of patients who have a CR or PR in the CNS, as determined by the Investigator according to RANO-BM criteria

SECONDARY OUTCOMES:
CNS CBR | from enrollment to progression or death (for any reason), assessed up to 24 months
  CNS clinical benefit rate (CBR) will be defined as the percentage of patients who experience a CR, PR or Stable Disease (SD) for at least 24 weeks.
Progression-free survival | Up to 2 years
  PFS will be defined as the time from the first dose of treatment to death or disease progression
Overall survival | Up to 2 years
  OS will be defined as the time from the first dose of treatment to death for any cause
First progression site | Up to 2 years
  The first lesion to progress
Safety as assessed by percentage of patients with any Adverse Event | Up to 2 years
  Adverse event according to NCI-CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Biyun wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China